CLINICAL TRIAL: NCT04233008
Title: Length of Cook Catheter Placement and Induction of Labor: a Randomized Controlled Trial
Brief Title: Length of Cook Catheter Placement and Induction of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Sarah E Little, Director of Clinical Research, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 54321
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Results first posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-05

CONDITIONS: Induction of Labor
Keywords: Maternal outcomes; Neonatal Outcomes

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 6 hour foley (Experimental): The participant will have a cook catheter inserted digitally or by direct visualization with a speculum with the uterine component of the balloon inflated to maximum 60mL. The catheter will be taped to the inner thigh with gentle traction. Participants will be started on hospital-based oxytocin protocol. The cook catheter will then be removed at 6 hours, determined by randomization. At that point health care providers will manage active labor.
  Interventions: Device: Foley catheter length
- 12 hour foley (No Intervention): The participant will have a cook catheter inserted digitally or by direct visualization with a speculum with the uterine component of the balloon inflated to maximum 60mL. The catheter will be taped to the inner thigh with gentle traction. Participants will be started on hospital-based oxytocin protocol. The cook catheter will then be removed at 12 hours, determined by randomization. At that point health care providers will manage active labor.

INTERVENTIONS:
Device: Foley catheter length — see arm description
  Arms: 6 hour foley

SUMMARY:
The goal of this study is to compare cook catheter placement for 6 vs. 12 hours to see if there is faster time to delivery for people admitted to labor and delivery undergoing induction of labor.

DETAILED DESCRIPTION:
Upon presentation to labor and delivery the participant will have a cook catheter inserted digitally or by direct visualization with a speculum. The uterine component of the balloon will be inflated to maximum 60mL. The catheter will be taped to the inner thigh with gentle traction. In both groups participants will be started on hospital-based oxytocin protocol. This protocol beings with 2 milliunits/min of oxytocin, increasing by 2 milliunits every 15 minutes until regular uterine contractions occur. The maximum dose of oxytocin is considered to be 30 milliunits. The cook catheter will then be removed at 6 vs. 12 hours based on randomization. At that point health care providers will manage active labor. Health care providers many perform amniotomy at any point during the induction process with recommendation for amniotomy with cervix more than 4cm dilated. Labor interventions are at the discretion of the healthcare provider. The participants will have continuous fetal monitoring throughout their induction, labor and delivery. Need for operative delivery or cesarean section will be at the discretion of the health provider.

ELIGIBILITY:
Inclusion Criteria: Women undergoing cervical ripening for labor induction at term (37-41 6/7 weeks) with a singleton gestation in cephalic presentation. Women will need to have a bishop score <6 or cervical dilation <2cm with intact membranes to be included.

Exclusion Criteria:

* Non English speaking
* Contraindications to vaginal delivery
* Prior cesarean section

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women only
Enrollment: 178 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Little, MD, Principal Investigator — Brigham and Women's Hospital, Harvard Medical School, Boston MA
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Research only shared within study staff

REFERENCES:
- [Background] Battarbee AN, Palatnik A, Peress DA, Grobman WA. Association of Early Amniotomy After Foley Balloon Catheter Ripening and Duration of Nulliparous Labor Induction. Obstet Gynecol. 2016 Sep;128(3):592-597. doi: 10.1097/AOG.0000000000001563. PMID 27500341
- [Background] Boulvain M, Kelly A, Lohse C, Stan C, Irion O. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2001;(4):CD001233. doi: 10.1002/14651858.CD001233. PMID 11687101
- [Background] Cromi A, Ghezzi F, Agosti M, Serati M, Uccella S, Arlant V, Bolis P. Is transcervical Foley catheter actually slower than prostaglandins in ripening the cervix? A randomized study. Am J Obstet Gynecol. 2011 Apr;204(4):338.e1-7. doi: 10.1016/j.ajog.2010.11.029. Epub 2011 Jan 26. PMID 21272849
- [Background] Hamilton BE, Martin JA, Osterman MJ, Curtin SC, Matthews TJ. Births: Final Data for 2014. Natl Vital Stat Rep. 2015 Dec;64(12):1-64. PMID 26727629
- [Background] Levine LD, Downes KL, Elovitz MA, Parry S, Sammel MD, Srinivas SK. Mechanical and Pharmacologic Methods of Labor Induction: A Randomized Controlled Trial. Obstet Gynecol. 2016 Dec;128(6):1357-1364. doi: 10.1097/AOG.0000000000001778. PMID 27824758
- [Derived] Lassey SC, Haber HR, Kanbergs A, Robinson JN, Little SE. Six versus twelve hours of single-balloon catheter placement with oxytocin administration for labor induction: a randomized controlled trial. Am J Obstet Gynecol. 2021 Jun;224(6):611.e1-611.e8. doi: 10.1016/j.ajog.2021.03.021. Epub 2021 Mar 23. PMID 33771496

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 6 Hour Foley | 12 Hour Foley
Started | 89 | 89
Completed | 89 | 89
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 6 Hour Foley: Foley for up to 6 hours
- 12 Hour Foley: Foley up to 12 hours
- Total: Total of all reporting groups
Arm/Group | 6 Hour Foley | 12 Hour Foley | Total
Number analyzed (Participants) | 89 | 88 | 177
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31.2 [28.4 to 33.1] | 31.4 [29 to 36.1] | 31.3 [28.6 to 34.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 88 | 177
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: white | 43 | 52 | 95
  Race/Ethnicity: Latinx | 20 | 12 | 32
  Race/Ethnicity: Black | 16 | 18 | 34
  Race/Ethnicity: Asian | 8 | 6 | 14
  Race/Ethnicity: Other | 2 | 0 | 2
Nulliparous [Count of Participants; unit: Participants] | 71 | 68 | 139
BMI [Median (Inter-Quartile Range); unit: kg/m2] | 30.1 [26.4 to 34.1] | 31.8 [27.5 to 36] | 31.0 [27.0 to 35.1]
Gestational Age [Median (Inter-Quartile Range); unit: Weeks] | 39 [38.3 to 39.7] | 39 [37.7 to 39.1] | 39 [37.2 to 39.4]
Bishop score at randomization [Median (Inter-Quartile Range); unit: units on a scale] — Scale 0-12, higher is more favorable cervix for induction
  units on a scale | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
Birthweight (g) [Median (Inter-Quartile Range); unit: grams] | 3200 [2905 to 3600] | 3149 [2797 to 3512] | 3175 [2851 to 3556]

OUTCOME MEASURES:

1. Primary Outcome: Time to Delivery
Description: Time to delivery
Time Frame: Assessed following delivery (delivery day, day 0)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | 6 Hour Foley | 12 Hour Foley
Number analyzed (Participants) | 89 | 88
hours | 19.2 [13.9 to 28] | 24.3 [15.6 to 32]
Statistical Analysis 1: Comparison: 6 Hour Foley vs 12 Hour Foley; Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Cesarean Delivery Rate
Description: Cesarean delivery rate
Time Frame: Assessed following delivery (delivery day, day 0)
Measure: Count of Participants; unit: Participants
Arm/Group | 6 Hour Foley | 12 Hour Foley
Number analyzed (Participants) | 89 | 88
Participants | 17 | 25
Statistical Analysis 1: Comparison: 6 Hour Foley vs 12 Hour Foley; Test type: Superiority; p = 0.14, Chi-squared

3. Secondary Outcome: Time to Active Labor
Description: Time to reaching active labor (defined as 5cm)
Time Frame: Assessed following delivery (delivery day, day 0)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | 6 Hour Foley | 12 Hour Foley
Number analyzed (Participants) | 85 | 82
hours | 10.5 [8.1 to 16.2] | 15.9 [10.7 to 23]
Statistical Analysis 1: Comparison: 6 Hour Foley vs 12 Hour Foley; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Delivery Within 12 Hours
Description: The number of women in each group who deliver within 12 hours
Time Frame: Assessed following delivery (delivery day, day 0)
Measure: Count of Participants; unit: Participants
Arm/Group | 6 Hour Foley | 12 Hour Foley
Number analyzed (Participants) | 89 | 88
Participants | 14 | 9
Statistical Analysis 1: Comparison: 6 Hour Foley vs 12 Hour Foley; Test type: Superiority; p = 0.39, Chi-squared

5. Secondary Outcome: Delivery Within 24 Hours
Description: The number of women in each group who deliver within 24 hours
Time Frame: Assessed following delivery (delivery day, day 0)
Measure: Count of Participants; unit: Participants
Arm/Group | 6 Hour Foley | 12 Hour Foley
Number analyzed (Participants) | 89 | 88
Participants | 60 | 42
Statistical Analysis 1: Comparison: 6 Hour Foley vs 12 Hour Foley; Test type: Superiority; p < 0.01, Chi-squared

6. Secondary Outcome: Maternal Length of Stay
Description: Length of hospital stay from start of induction to postpartum discharge
Time Frame: Assessed at end of study period (week 4)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | 6 Hour Foley | 12 Hour Foley
Number analyzed (Participants) | 89 | 88
days | 2 [2 to 3] | 2 [2 to 3.5]

7. Secondary Outcome: Indication for Cesarean Delivery
Description: Number of Patient with Indication for Cesarean Delivery
Time Frame: Assessed following delivery (delivery day, day 0)
Measure: Count of Participants; unit: Participants
Arm/Group | 6 Hour Foley | 12 Hour Foley
Number analyzed (Participants) | 17 | 25
Participants | 10 | 11
Statistical Analysis 1: Comparison: 6 Hour Foley vs 12 Hour Foley; Test type: Superiority; p = 0.8, Chi-squared

8. Secondary Outcome: Maternal Complications
Description: Estimated blood loss, blood transfusion, higher order laceration, endometritis, wound infection, venous thromboembolism, hysterectomy, ICU admission, maternal death
Time Frame: Assessed at end of study period (week 4)
Measure: Count of Participants; unit: Participants
Arm/Group | 6 Hour Foley | 12 Hour Foley
Number analyzed (Participants) | 89 | 88
Participants
  Postpartum hemorrage | 7 | 8
  Higher order laceration | 7 | 2
  Wound infection | 1 | 1
  Endometritis | 1 | 1
  chorioamnionitis | 13 | 11

9. Secondary Outcome: Neonatal Complications
Description: culture-proven neonatal sepsis, neonatal blood transfusion, hypoxic-ischemic encephalopathy, intraventricular hemorrhage grade 3 or 4, or therapeutic hypothermia
Time Frame: Assessed at end of study period (week 4)
Measure: Count of Participants; unit: Participants
Arm/Group | 6 Hour Foley | 12 Hour Foley
Number analyzed (Participants) | 89 | 88
Participants | 0 | 0

10. Secondary Outcome: NICU Admission
Description: Number of infants admitted to NICU
Time Frame: Assessed at end of study period (week 4)
Measure: Count of Participants; unit: Participants
Arm/Group | 6 Hour Foley | 12 Hour Foley
Number analyzed (Participants) | 89 | 88
Participants | 9 | 6

11. Secondary Outcome: NICU Admission >48 Hours
Description: Number of infants admitted to NICU for >48 hours
Time Frame: Assessed at end of study period (week 4)
Measure: Count of Participants; unit: Participants
Arm/Group | 6 Hour Foley | 12 Hour Foley
Number analyzed (Participants) | 89 | 88
Participants | 4 | 2

12. Secondary Outcome: Neonatal Length of Stay
Description: Days of hospital stay
Time Frame: Assessed at end of study period (week 4)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | 6 Hour Foley | 12 Hour Foley
Number analyzed (Participants) | 89 | 88
days | 2 [2 to 4] | 2 [2 to 4]

ADVERSE EVENTS:
Time Frame: Up to 4 week postpartum
Groups:
- 6 Hour Foley - Mothers; 6 Hour Foley - Neonates: The participant will have a cook catheter inserted digitally or by direct visualization with a speculum with the uterine component of the balloon inflated to maximum 60mL. The catheter will be taped to the inner thigh with gentle traction. Participants will be started on hospital-based oxytocin protocol. The cook catheter will then be removed at 6 hours, determined by randomization. At that point health care providers will manage active labor.
  Foley catheter length: see arm description
- 12 Hour Foley - Mothers; 12 Hour Foley - Neonates: The participant will have a cook catheter inserted digitally or by direct visualization with a speculum with the uterine component of the balloon inflated to maximum 60mL. The catheter will be taped to the inner thigh with gentle traction. Participants will be started on hospital-based oxytocin protocol. The cook catheter will then be removed at 12 hours, determined by randomization. At that point health care providers will manage active labor.
Arm/Group | 6 Hour Foley - Mothers | 12 Hour Foley - Mothers | 6 Hour Foley - Neonates | 12 Hour Foley - Neonates
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/89 | 0/89 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/89 | 0/89 | 0/89
Other Adverse Events (participants affected / at risk) | 0/89 | 0/89 | 0/89 | 0/89

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT04233008/Prot_SAP_000.pdf